CLINICAL TRIAL: NCT00000526
Title: Cardiac Arrhythmia Suppression Trial (CAST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 45
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Death, Sudden, Cardiac; Heart Arrest; Heart Diseases; Myocardial Infarction; Myocardial Ischemia; Ventricular Arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Death, Sudden, Cardiac; Heart Arrest; Heart Diseases; Myocardial Infarction; Myocardial Ischemia | interventions — Encainide; Flecainide; Moricizine

INTERVENTIONS:
Drug: encainide
Drug: flecainide
Drug: moricizine

SUMMARY:
To determine whether drug treatment of asymptomatic ventricular arrhythmias in post-myocardial infarction patients reduced the incidence of sudden cardiac death and total mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Each year over 400,000 people in the United States die suddenly of coronary heart disease. The majority have known coronary heart disease. Of these, the post-myocardial infarction population constitutes a large proportion. About 8 to 15 percent of patients who recover from an acute myocardial infarction die in the subsequent year. Half of these deaths are usually sudden, presumably due to arrhythmia. Advanced age, poor ventricular function, and presence of ventricular arrhythmias can identify post-MI patients at high risk of sudden cardiac death and all-cause mortality.

A number of clinical trials have evaluated whether acute or chronic anti-arrhythmic drug therapy can reduce mortality in post-MI patients. Of these, only the use of acute intravenous and long-term beta-blockers, independently and in combination, had been shown to reduce mortality. However, beta-blockers have many actions in addition to being anti-arrhythmic agents and it is possible that these other effects may have been particularly important in prolonging life.

None of the clinical trials of other antiarrhythmic drugs had shown significant benefits from treatment, and a number had even failed to show a positive trend. It was certainly possible that treatment of ventricular premature depolarizations, in itself, did not lead to a reduction in mortality, or even sudden death. The studies that had been done, however, had not adequately addressed the issue. Most of the studies were small and did not select patients on the basis of frequent ectopic beats. Moreover, appropriate drugs in optimal doses may not have been used, and adverse effects may well have outweighed any potential benefit. Poor compliance, perhaps due to adverse effects, may also have limited the opportunity for a beneficial outcome.

In an effort to address some of these points, the National Heart, Lung, and Blood Institute initiated the Cardiac Arrhythmia Pilot Study in 1982. The objectives were to assess: whether post-MI patients with documented ventricular arrhythmia could be identified and enrolled into a double-blind clinical trial; whether one or more drugs could be found to effectively and safely reduce ventricular premature depolarizations over a one-year period; whether dose-adjustment could be carried out, using ambulatory ECG's; and whether good patient compliance could be maintained. The Cardiac Arrhythmia Pilot Study, which enrolled 500 patients, evaluated four active drugs (encainide, ethmozine, flecainide, imipramine) against placebo. The study was too small to determine whether any of these drugs had an effect on mortality or major morbidity. The study was completed in July 1986.

The pilot study demonstrated that patient recruitment was feasible, that dose-adjustment could be accomplished, and that good compliance to the protocol could be achieved. Because of the encouraging results of the pilot study, the NHLBI conducted a full-scale trial.

DESIGN NARRATIVE:

Randomized, double-blind. Enrollment began in June 1987 when twenty-seven clinical centers began to randomize 4,400 post-myocardial infarction patients to placebo or treatment with encainide, flecainide, or moricizine. Prior to actual randomization, there was an open-label titration period to identify patients who responded to treatment. A total of 1,727 patients who responded were randomized: 1,455 to encainide, flecainide, or placebo, and 272 to moricizine or placebo. In April 1989, encainide and flecainide were discontinued because of increased total mortality and sudden arrhythmic death. CAST continued to compare moricizine to placebo in 1,300 patients for 18 months until August 1991 when the moricizine portion of the trial was stopped early because of excess deaths. The primary outcome variable in the full-scale trial was sudden cardiac death, with total mortality a secondary endpoint. Data analysis continued through March 1998.

ELIGIBILITY:
Men and women with ventricular premature depolarization six days to two years after the start of myocardial infarction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1986-08; Study Completion 1998-03

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Hallstrom — University of Washington

REFERENCES:
- [Background] Pratt CM, Moye LA. The cardiac arrhythmia suppression trial. Casting suppression in a different light. Circulation. 1995 Jan 1;91(1):245-7. doi: 10.1161/01.cir.91.1.245. No abstract available. PMID 7805210
- [Background] el-Sherif N, Denes P, Katz R, Capone R, Mitchell LB, Carlson M, Reynolds-Haertle R. Definition of the best prediction criteria of the time domain signal-averaged electrocardiogram for serious arrhythmic events in the postinfarction period. The Cardiac Arrhythmia Suppression Trial/Signal-Averaged Electrocardiogram (CAST/SAECG) Substudy Investigators. J Am Coll Cardiol. 1995 Mar 15;25(4):908-14. doi: 10.1016/0735-1097(94)00504-j. PMID 7884096
- [Background] Cardiac Arrhythmia Suppression Trial (CAST) Investigators. Preliminary report: effect of encainide and flecainide on mortality in a randomized trial of arrhythmia suppression after myocardial infarction. N Engl J Med. 1989 Aug 10;321(6):406-12. doi: 10.1056/NEJM198908103210629. PMID 2473403
- [Background] Bigger JT Jr. The events surrounding the removal of encainide and flecainide from the Cardiac Arrhythmia Suppression Trial (CAST) and why CAST is continuing with moricizine. J Am Coll Cardiol. 1990 Jan;15(1):243-5. doi: 10.1016/0735-1097(90)90209-8. No abstract available. PMID 2104884
- [Background] Morganroth J, Bigger JT Jr, Anderson JL. Treatment of ventricular arrhythmias by United States cardiologists: a survey before the Cardiac Arrhythmia Suppression Trial results were available. Am J Cardiol. 1990 Jan 1;65(1):40-8. doi: 10.1016/0002-9149(90)90023-t. PMID 1688481
- [Background] Pratt CM, Moye LA. The Cardiac Arrhythmia Suppression Trial: background, interim results and implications. Am J Cardiol. 1990 Jan 16;65(4):20B-29B. doi: 10.1016/0002-9149(90)91287-g. PMID 2105049
- [Background] Pratt CM. The Cardiac Arrhythmia Suppression Trial. Introduction: The aftermath of the CAST--a reconsideration of traditional concepts. Am J Cardiol. 1990 Jan 16;65(4):1B-2B. doi: 10.1016/0002-9149(90)91283-c. No abstract available. PMID 2404392
- [Background] Pratt CM, Brater DC, Harrell FE Jr, Kowey PR, Leier CV, Lowenthal DT, Messerli F, Packer M, Pritchett EL, Ruskin JN. Clinical and regulatory implications of the Cardiac Arrhythmia Suppression Trial. Am J Cardiol. 1990 Jan 1;65(1):103-5. doi: 10.1016/0002-9149(90)90034-x. No abstract available. PMID 1688479
- [Background] Pratt CM, Moye L. The cardiac arrhythmia suppression trial: implications for antiarrhythmic drug development. J Clin Pharmacol. 1990 Nov;30(11):967-74. doi: 10.1002/j.1552-4604.1990.tb03580.x. No abstract available. PMID 2122983
- [Background] Bigger JT Jr. Implications of the Cardiac Arrhythmia Suppression Trial for antiarrhythmic drug treatment. Am J Cardiol. 1990 Feb 20;65(8):3D-10D; discussion 68D-71D. doi: 10.1016/0002-9149(90)91410-8. PMID 2106253
- [Background] Morganroth J, Bigger JT Jr. Pharmacologic management of ventricular arrhythmias after the cardiac arrhythmia suppression trial. Am J Cardiol. 1990 Jun 15;65(22):1497-503. doi: 10.1016/0002-9149(90)91362-a. No abstract available. PMID 2091621
- [Background] Echt DS, Liebson PR, Mitchell LB, Peters RW, Obias-Manno D, Barker AH, Arensberg D, Baker A, Friedman L, Greene HL, et al. Mortality and morbidity in patients receiving encainide, flecainide, or placebo. The Cardiac Arrhythmia Suppression Trial. N Engl J Med. 1991 Mar 21;324(12):781-8. doi: 10.1056/NEJM199103213241201. PMID 1900101
- [Background] Epstein AE, Bigger JT Jr, Wyse DG, Romhilt DW, Reynolds-Haertle RA, Hallstrom AP. Events in the Cardiac Arrhythmia Suppression Trial (CAST): mortality in the entire population enrolled. J Am Coll Cardiol. 1991 Jul;18(1):14-9. doi: 10.1016/s0735-1097(10)80210-4. PMID 1904891
- [Background] Wyse DG, Hallstrom A, McBride R, Cohen JD, Steinberg JS, Mahmarian J. Events in the Cardiac Arrhythmia Suppression Trial (CAST): mortality in patients surviving open label titration but not randomized to double-blind therapy. J Am Coll Cardiol. 1991 Jul;18(1):20-8. doi: 10.1016/s0735-1097(10)80211-6. PMID 1904892
- [Background] Hallstrom AP, Verter J, Friedman L. Randomizing responders. Cardiac Arrhythmia Suppression Trial (CAST) investigators. Control Clin Trials. 1991 Aug;12(4):486-503. doi: 10.1016/0197-2456(91)90009-b. PMID 1657526
- [Background] Denes P, Gillis AM, Pawitan Y, Kammerling JM, Wilhelmsen L, Salerno DM. Prevalence, characteristics and significance of ventricular premature complexes and ventricular tachycardia detected by 24-hour continuous electrocardiographic recording in the Cardiac Arrhythmia Suppression Trial. CAST Investigators. Am J Cardiol. 1991 Oct 1;68(9):887-96. doi: 10.1016/0002-9149(91)90404-9. PMID 1718158
- [Background] Capone RJ, Pawitan Y, el-Sherif N, Geraci TS, Handshaw K, Morganroth J, Schlant RC, Waldo AL. Events in the cardiac arrhythmia suppression trial: baseline predictors of mortality in placebo-treated patients. J Am Coll Cardiol. 1991 Nov 15;18(6):1434-8. doi: 10.1016/0735-1097(91)90671-u. PMID 1939943
- [Background] Hallstrom AP, Greene HL, Huther ML. The healthy responder phenomenon in non-randomized clinical trials. CAST Investigators. Stat Med. 1991 Oct;10(10):1621-31. doi: 10.1002/sim.4780101013. PMID 1947517
- [Background] Greene HL, Roden DM, Katz RJ, Woosley RL, Salerno DM, Henthorn RW. The Cardiac Arrhythmia Suppression Trial: first CAST ... then CAST-II. J Am Coll Cardiol. 1992 Apr;19(5):894-8. doi: 10.1016/0735-1097(92)90267-q. PMID 1552108
- [Background] Cardiac Arrhythmia Suppression Trial II Investigators. Effect of the antiarrhythmic agent moricizine on survival after myocardial infarction. N Engl J Med. 1992 Jul 23;327(4):227-33. doi: 10.1056/NEJM199207233270403. PMID 1377359
- [Background] Akiyama T, Pawitan Y, Campbell WB, Papa L, Barker AH, Rubbert P, Friedman L, Keller M, Josephson RA. Effects of advancing age on the efficacy and side effects of antiarrhythmic drugs in post-myocardial infarction patients with ventricular arrhythmias. The CAST Investigators. J Am Geriatr Soc. 1992 Jul;40(7):666-72. doi: 10.1111/j.1532-5415.1992.tb01957.x. PMID 1607582
- [Background] Shea S, Bigger JT Jr, Campion J, Fleiss JL, Rolnitzky LM, Schron E, Gorkin L, Handshaw K, Kinney MR, Branyon M. Enrollment in clinical trials: institutional factors affecting enrollment in the cardiac arrhythmia suppression trial (CAST). Control Clin Trials. 1992 Dec;13(6):466-86. doi: 10.1016/0197-2456(92)90204-d. PMID 1334819
- [Background] Willund I, Gorkin L, Pawitan Y, Schron E, Schoenberger J, Jared LL, Shumaker S. Methods for assessing quality of life in the cardiac arrhythmia suppression trial (CAST). Qual Life Res. 1992 Jun;1(3):187-201. doi: 10.1007/BF00635618. PMID 1301128
- [Background] Reynolds-Haertle RA, McBride R. Single vs. double data entry in CAST. Control Clin Trials. 1992 Dec;13(6):487-94. doi: 10.1016/0197-2456(92)90205-e. PMID 1334820
- [Background] Gorkin L, Schron EB, Brooks MM, Wiklund I, Kellen J, Verter J, Schoenberger JA, Pawitan Y, Morris M, Shumaker S. Psychosocial predictors of mortality in the Cardiac Arrhythmia Suppression Trial-1 (CAST-1). Am J Cardiol. 1993 Feb 1;71(4):263-7. doi: 10.1016/0002-9149(93)90788-e. PMID 8427165
- [Background] Peters RW, Zoble RG, Liebson PR, Pawitan Y, Brooks MM, Proschan M. Identification of a secondary peak in myocardial infarction onset 11 to 12 hours after awakening: the Cardiac Arrhythmia Suppression Trial (CAST) experience. J Am Coll Cardiol. 1993 Oct;22(4):998-1003. doi: 10.1016/0735-1097(93)90408-s. PMID 8409074
- [Background] Epstein AE, Hallstrom AP, Rogers WJ, Liebson PR, Seals AA, Anderson JL, Cohen JD, Capone RJ, Wyse DG. Mortality following ventricular arrhythmia suppression by encainide, flecainide, and moricizine after myocardial infarction. The original design concept of the Cardiac Arrhythmia Suppression Trial (CAST). JAMA. 1993 Nov 24;270(20):2451-5. PMID 8230622
- [Background] Friedman LM, Bristow JD, Hallstrom A, Schron E, Proschan M, Verter J, DeMets D, Fisch C, Nies AS, Ruskin J, et al. Data monitoring in the cardiac arrhythmia suppression trial. Online J Curr Clin Trials. 1993 Jul 31;Doc No 79:[5870 words; 53 paragraphs]. doi: 10.1007/0-387-30107-0_18. PMID 8306012
- [Background] Peters RW, Mitchell LB, Brooks MM, Echt DS, Barker AH, Capone R, Liebson PR, Greene HL. Circadian pattern of arrhythmic death in patients receiving encainide, flecainide or moricizine in the Cardiac Arrhythmia Suppression Trial (CAST). J Am Coll Cardiol. 1994 Feb;23(2):283-9. doi: 10.1016/0735-1097(94)90408-1. PMID 8294678
- [Background] Wyse DG, Morganroth J, Ledingham R, Denes P, Hallstrom A, Mitchell LB, Epstein AE, Woosley RL, Capone R. New insights into the definition and meaning of proarrhythmia during initiation of antiarrhythmic drug therapy from the Cardiac Arrhythmia Suppression Trial and its pilot study. The CAST and CAPS Investigators. J Am Coll Cardiol. 1994 Apr;23(5):1130-40. doi: 10.1016/0735-1097(94)90601-7. PMID 8144779
- [Background] Hochman JS, Brooks MM, Morris M, Ahmad T. Prognostic significance of left ventricular aneurysm in the Cardiac Arrhythmia Suppression Trial (CAST) population. Am Heart J. 1994 Apr;127(4 Pt 1):824-32. doi: 10.1016/0002-8703(94)90549-5. PMID 8154420
- [Background] Denes P, el-Sherif N, Katz R, Capone R, Carlson M, Mitchell LB, Ledingham R. Prognostic significance of signal-averaged electrocardiogram after thrombolytic therapy and/or angioplasty during acute myocardial infarction (CAST substudy). Cardiac Arrhythmia Suppression Trial (CAST) SAECG Substudy Investigators. Am J Cardiol. 1994 Aug 1;74(3):216-20. doi: 10.1016/0002-9149(94)90359-x. PMID 8037124
- [Background] Anderson JL, Platia EV, Hallstrom A, Henthorn RW, Buckingham TA, Carlson MD, Carson PE. Interaction of baseline characteristics with the hazard of encainide, flecainide, and moricizine therapy in patients with myocardial infarction. A possible explanation for increased mortality in the Cardiac Arrhythmia Suppression Trial (CAST). Circulation. 1994 Dec;90(6):2843-52. doi: 10.1161/01.cir.90.6.2843. PMID 7994829
- [Background] Brooks MM, Gorkin L, Schron EB, Wiklund I, Campion J, Ledingham RB. Moricizine and quality of life in the Cardiac Arrhythmia Suppression Trial II (CAST II). Control Clin Trials. 1994 Dec;15(6):437-49. doi: 10.1016/0197-2456(94)90002-7. PMID 7851106
- [Background] Kennedy HL, Brooks MM, Barker AH, Bergstrand R, Huther ML, Beanlands DS, Bigger JT, Goldstein S. Beta-blocker therapy in the Cardiac Arrhythmia Suppression Trial. CAST Investigators. Am J Cardiol. 1994 Oct 1;74(7):674-80. doi: 10.1016/0002-9149(94)90308-5. PMID 7942525
- [Background] Hallstrom A, Pratt CM, Greene HL, Huther M, Gottlieb S, DeMaria A, Young JB. Relations between heart failure, ejection fraction, arrhythmia suppression and mortality: analysis of the Cardiac Arrhythmia Suppression Trial. J Am Coll Cardiol. 1995 May;25(6):1250-7. doi: 10.1016/0735-1097(94)00553-3. PMID 7722117
- [Background] A symposium: the cardiac arrhythmia suppression trial--does it alter our concepts of and approaches to ventricular arrhythmias? Woodland, Texas, August 9, 1989. Am J Cardiol. 1990 Jan 16;65(4):1B-42B. No abstract available. PMID 2404393
- [Background] Akiyama T, Pawitan Y, Greenberg H, Kuo CS, Reynolds-Haertle RA. Increased risk of death and cardiac arrest from encainide and flecainide in patients after non-Q-wave acute myocardial infarction in the Cardiac Arrhythmia Suppression Trial. CAST Investigators. Am J Cardiol. 1991 Dec 15;68(17):1551-5. doi: 10.1016/0002-9149(91)90308-8. PMID 1720917
- [Background] Hallstrom AP, Anderson JL, Carlson M, Davies R, Greene HL, Kammerling JM, Romhilt DW, Duff HJ, Huther M. Time to arrhythmic, ischemic, and heart failure events: exploratory analyses to elucidate mechanisms of adverse drug effects in the Cardiac Arrhythmia Suppression Trial. Am Heart J. 1995 Jul;130(1):71-9. doi: 10.1016/0002-8703(95)90238-4. PMID 7611126
- [Background] Friedmann E, Thomas SA. Pet ownership, social support, and one-year survival after acute myocardial infarction in the Cardiac Arrhythmia Suppression Trial (CAST). Am J Cardiol. 1995 Dec 15;76(17):1213-7. doi: 10.1016/s0002-9149(99)80343-9. PMID 7502998
- [Background] Roose SP, Glassman AH. Antidepressant choice in the patient with cardiac disease: lessons from the Cardiac Arrhythmia Suppression Trial (CAST) studies. J Clin Psychiatry. 1994 Sep;55 Suppl A:83-7; discussion 88-9, 98-100. PMID 7961547
- [Background] Josephson RA, Chahine RA, Morganroth J, Anderson J, Waldo A, Hallstrom A. Prediction of cardiac death in patients with a very low ejection fraction after myocardial infarction: a Cardiac Arrhythmia Suppression Trial (CAST) study. Am Heart J. 1995 Oct;130(4):685-91. doi: 10.1016/0002-8703(95)90064-0. PMID 7572573
- [Background] Peters RW, Brooks MM, Todd L, Liebson PR, Wilhelmsen L. Smoking cessation and arrhythmic death: the CAST experience. The Cardiac Arrhythmia Suppression Trial (CAST) Investigators. J Am Coll Cardiol. 1995 Nov 1;26(5):1287-92. doi: 10.1016/0735-1097(95)00328-2. PMID 7594045
- [Background] Kellen JC, Ettinger A, Todd L, Brezsnyak ML, Campion J, McBride R, Thomas S, Corum J, Schron E. The Cardiac Arrhythmia Suppression Trial: Implications for nursing practice. Am J Crit Care. 1996 Jan;5(1):19-25. PMID 8680488
- [Background] Schron EB, Brooks MM, Gorkin L, Kellen JC, Morris M, Campion J, Shumaker SA, Corum J. Relation of sociodemographic, clinical, and quality-of-life variables to adherence in the cardiac arrhythmia suppression trial. Cardiovasc Nurs. 1996 Mar-Apr;32(2):1-6. PMID 8697488
- [Background] Peters RW, Brooks MM, Zoble RG, Liebson PR, Seals AA. Chronobiology of acute myocardial infarction: cardiac arrhythmia suppression trial (CAST) experience. Am J Cardiol. 1996 Dec 1;78(11):1198-201. doi: 10.1016/s0002-9149(96)00595-4. PMID 8960574
- [Background] Goldstein S, Zoble RG, Akiyama T, Cohen JD, Lancaster S, Liebson PR, Rapaport E, Goldberg AD, Peters RW, Gillis AM. Relation of circadian ventricular ectopic activity to cardiac mortality. CAST Investigators. Am J Cardiol. 1996 Oct 15;78(8):881-5. doi: 10.1016/s0002-9149(96)00461-4. PMID 8888659
- [Background] Obias-Manno D, Friedmann E, Brooks MM, Thomas SA, Haakenson C, Morris M, Wimbush F, Somelofski C, Goldner F. Adherence and arrhythmic mortality in the cardiac arrhythmia suppression trial (CAST). Ann Epidemiol. 1996 Mar;6(2):93-101. doi: 10.1016/1047-2797(95)00134-4. PMID 8775589
- [Background] Gorkin L, Schron EB, Handshaw K, Shea S, Kinney MR, Branyon M, Campion J, Bigger JT Jr, Sylvia SC, Duggan J, Stylianou M, Lancaster S, Ahern DK, Follick MJ. Clinical trial enrollers vs. nonenrollers: the Cardiac Arrhythmia Suppression Trial (CAST) Recruitment and Enrollment Assessment in Clinical Trials (REACT) project. Control Clin Trials. 1996 Feb;17(1):46-59. doi: 10.1016/0197-2456(95)00089-5. PMID 8721801
- [Background] Anderson JL, Karagounis LA, Stein KM, Moreno FL, Ledingham R, Hallstrom A. Predictive value for future arrhythmic events of fractal dimension, a measure of time clustering of ventricular premature complexes, after myocardial infarction. CAST Investigators. Cardia Arrhythmia Suppression Trial. J Am Coll Cardiol. 1997 Jul;30(1):226-32. doi: 10.1016/s0735-1097(97)00108-3. PMID 9207646
- [Background] Thomas SA, Friedmann E, Wimbush F, Schron E. Psychological factors and survival in the cardiac arrhythmia suppression trial (CAST): a reexamination. Am J Crit Care. 1997 Mar;6(2):116-26. PMID 9172848
- [Background] Shumaker SA, Brooks MM, Schron EB, Hale C, Kellen JC, Inkster M, Wimbush FB, Wiklund I, Morris M. Gender differences in health-related quality of life among postmyocardial infarction patients: brief report. CAST Investigators. Cardiac Arrhythmia Suppression Trials. Womens Health. 1997 Spring;3(1):53-60. PMID 9106370
- [Background] Every NR, Hlatky MA, McDonald KM, Weaver WD, Hallstrom AP. Estimating the proportion of post-myocardial infarction patients who may benefit from prophylactic implantable defibrillator placement from analysis of the CAST registry. Cardiac Arrhythmia Suppression Trial. Am J Cardiol. 1998 Sep 1;82(5):683-5, A8. doi: 10.1016/s0002-9149(98)00417-2. PMID 9732904
- [Background] Hallstrom A, Friedman L, Denes P, Rizo-Patron C, Morris M; CAST Investigators; AVID Investigators. Do arrhythmia patients improve survival by participating in randomized clinical trials? Observations from the Cardiac Arrhythmia Suppression Trial (CAST)and the Antiarrhythmics Versus Implantable Defibrillators Trial (AVID). Control Clin Trials. 2003 Jun;24(3):341-52. doi: 10.1016/s0197-2456(03)00002-3. PMID 12757998
- [Background] Ruskin JN. The cardiac arrhythmia suppression trial (CAST). N Engl J Med. 1989 Aug 10;321(6):386-8. doi: 10.1056/NEJM198908103210608. No abstract available. PMID 2501683
- [Background] Goldstein S, Brooks MM, Ledingham R, Kennedy HL, Epstein AE, Pawitan Y, Bigger JT. Association between ease of suppression of ventricular arrhythmia and survival. Circulation. 1995 Jan 1;91(1):79-83. doi: 10.1161/01.cir.91.1.79. PMID 7805221
- Available data/document: Individual Participant Data Set: CAST — http://biolincc.nhlbi.nih.gov/studies/cast/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/cast/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/cast/